CLINICAL TRIAL: NCT04647032
Title: Enhancing Cognitive Control in Mild Cognitive Impairment Via Non-invasive Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132026a; R21AG062395 (NIH)
Record Dates: First submitted 2020-11-10; First posted 2020-11-30 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Theta Stimulation Group (Experimental): This group will receive 6 Hz (theta) stimulation
  Interventions: Device: Transcranial alternating current stimulation
- Delta Stimulation Group (Active Comparator): This group will receive 1 Hz (delta) stimulation
  Interventions: Device: Transcranial alternating current stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation — Transcranial alternating current stimulation (tACS) will be applied across the prefrontal cortex near electrodes coordinates AF3/AF4

SUMMARY:
The overall goal of this project is to improve cognitive control abilities in adults with mild cognitive impairment (MCI) through a form of non-invasive brain stimulation, transcranial alternating current stimulation (tACS).

DETAILED DESCRIPTION:
30 older adults aged 60-80 years with md-aMCI were randomized to 8 sessions of transcranial alternating current stimulation (tACS) with simultaneous cognitive control training (CCT). The intervention took place within the participant's home without direct researcher assistance. Half of the participants received prefrontal theta tACS during CCT and the other half received control tACS. Outcomes were assessed pre and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Grade 12 or more education
* Normal or corrected to normal vision and hearing
* Ability to complete cognitive tasks
* Ability to cooperate and comply with all study procedures
* Ability to tolerate tACS
* Montreal Cognitive Assessment score: 17-28
* -1 z-score on immediate memory, delayed memory, fluency, processing speed, or task switch
* Self-reported memory complaint

Exclusion Criteria:

* Neurological or psychiatric disorders other than mild cognitive impairment
* Receiving investigational medications or have participated in a trial with investigational medications within last 30 days
* Family history of epilepsy
* Implanted electronic devices (e.g., pacemaker)
* Prior head trauma
* Pregnant
* IQ < 80
* Taking cholinesterase inhibitory, memantine, or psychotropic medication
* Taking anti-depressants or anti-anxiety medication
* Color blind
* Substance abuse
* Glaucoma
* Macular degeneration
* Amblyopia (lazy eye)
* Strabismus (crossed eyes)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Zanto, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The dataset includes self-reported information, behavioral and electrophysiological data. The final dataset will be stripped of identifiers prior to release for sharing, thereby anonymizing the data. We will make the anonymized data available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to attempt to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. This will be in accordance with human subject regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after the results have been determined and the study researchers are unblinded. The data will be available indefinitely upon request.
Access Criteria: Contact PI.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Started | 15 | 15
Completed | 14 | 13
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theta Stimulation Group | Delta Stimulation Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (6) | 70 (4) | 70 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Divided Attention [Mean (Standard Deviation); unit: difficulty level achieved] — Divided attention was assessed as the difficulty level achieved during perceptual discrimination performance while participants were engaged in the Akili AKL-T01 task. Population: Difficulty level is a continuous unitless quantity that relates to the difficulty of the task. Higher is better.
  difficulty level achieved | 8.01 (1.56) | 8.51 (1.65) | 8.27 (1.61)
Sustained Attention [Mean (Standard Deviation); unit: milliseconds] — Sustained attention was assessed via response times during the continuous performance task. Population: Response times to visual targets. Lower is better.
  milliseconds | 527 (108) | 432 (56) | 481 (82)
Working Memory [Mean (Standard Deviation); unit: number correct] — Working memory was assessed as the average maximum number correct from the ACE-X span tasks. Population: Number of items remembered. Higher is better.
  number correct | 6.13 (0.96) | 6.56 (0.81) | 6.34 (0.89)
Instrumental Activities of Daily Living [Mean (Standard Deviation); unit: score on a scale] — Population: Higher is better (max = 4)
  score on a scale | 3.92 (0.29) | 4 (0) | 3.96 (0.14)

OUTCOME MEASURES:

1. Primary Outcome: Divided Attention Performance
Description: Divided attention was assessed as the difficulty level achieved during perceptual discrimination performance while participants were engaged in the Akili AKL-T01 task. Higher is better.
Time Frame: Post-tACS (1-day follow-up), approximately 1 week after baseline
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: difficulty level acheived
Groups:
- Theta Stimulation Group: This group received 6 Hz (theta) stimulation
  Transcranial alternating current stimulation: Transcranial alternating current stimulation (tACS) was applied across the prefrontal cortex near electrodes coordinates AF3/AF4
- Delta Stimulation Group: This group received 1 Hz (delta) stimulation
  Transcranial alternating current stimulation: Transcranial alternating current stimulation (tACS) was applied across the prefrontal cortex near electrodes coordinates AF3/AF4
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Number analyzed (Participants) | 14 | 13
difficulty level acheived | 9.29 (2.83) | 9.31 (2.40)

2. Primary Outcome: Divided Attention Performance
Description: as for outcome 1
Time Frame: Post-tACS (1-month follow-up), approximately 1 month after baseline
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: difficulty level acheived
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Number analyzed (Participants) | 14 | 13
difficulty level acheived | 10.10 (1.40) | 10.67 (1.18)

3. Primary Outcome: Sustained Attention Performance
Description: Sustained attention was assessed via response times to visual targets during the continuous performance task. Lower is better.
Time Frame: Post-tACS (1-day follow-up), approximately 1 week after baseline
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Number analyzed (Participants) | 14 | 13
milliseconds | 436 (73) | 416 (60)

4. Primary Outcome: Sustained Attention Performance
Description: as for outcome 3
Time Frame: Post-tACS (1-month follow-up), approximately 1 month after baseline
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Number analyzed (Participants) | 14 | 13
milliseconds | 428 (64) | 395 (49)

5. Primary Outcome: Working Memory Performance
Description: Working memory was assessed as the average maximum number correct from the ACE-X span tasks - memory for order of illuminated squares.
Time Frame: Post-tACS (1-day follow-up), approximately 1 week after baseline
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Number analyzed (Participants) | 14 | 13
number correct | 6.09 (1.29) | 6.89 (0.78)

6. Primary Outcome: Working Memory Performance
Description: as for outcome 5
Time Frame: Post-tACS (1-month follow-up), approximately 1 month after baseline
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Number analyzed (Participants) | 14 | 13
number correct | 6.13 (1.15) | 6.50 (0.75)

7. Secondary Outcome: Instrumental Activities of Daily Living (IADL)
Description: Scores on the IADL will be assessed pre and post intervention. Higher scores are better (minimum = 0, maximum = 4).
Time Frame: Post-tACS (1-day follow-up), approximately 1 week after baseline
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Number analyzed (Participants) | 14 | 13
score on a scale | 3.92 (0.29) | 4 (0)

8. Secondary Outcome: Instrumental Activities of Daily Living (IADL)
Description: Scores on the IADL will be assessed pre and post intervention. Higher scores are better (minimum = 0, maximum = 4).
Time Frame: Post-tACS (1-month follow-up), approximately 1 month after baseline
Population: Only data from participants who completed the full protocol were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
Number analyzed (Participants) | 14 | 13
score on a scale | 4 (0) | 4 (0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Theta Stimulation Group | Delta Stimulation Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04647032/Prot_SAP_002.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04647032/ICF_001.pdf